CLINICAL TRIAL: NCT06631872
Title: Implementing Tele-prehabilitation Education Into Cancer Care Pathways
Brief Title: Implementing Surgery School Prehabilitation Using Telehealth
Acronym: STTARRS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Melbourne (Other)
Collaborators: Peter MacCallum Cancer Centre, Australia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 4.2 19/02/2025
Record Dates: First submitted 2024-09-15; First posted 2024-10-08 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2024-10

CONDITIONS: Adults Waiting to Undergo Lung Cancer or Major Abdominal, Open or Video Assisted Cancer Surgery

STUDY DESIGN:
Intervention Model Description: This is a two-arm, multicentre, comparative, assessor-blinded, randomised, controlled, hybrid (Type 1; examining both efficacy and feasibility) superiority trial that includes one sub-study.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Tele-prehabilitation intervention (Intervention Group) (Experimental): The Teleprehabilitaiton intervention (also known as Surgery School) is a one-off group based education session delivered online. Video presentations of 8-10 key prehabilitation education areas will be facilitated by a live clinician facilitator who will introduce the educational content and answer any questions. All standardised video presentations during the session will be made available to participants through an online password-protected video repository hosted on a video platform after the session and will be available until their surgery.
  Interventions: Behavioral: Tele-prehabilitation education session: Surgery School
- Usual care alone (Control Group) (Active Comparator): Participants allocated to the control group will receive usual care according to their health care team, which may consist of advice on smoking cessation, reduction of alcohol intake, nutritional counselling and medical optimisation in preoperative anaesthetic clinic visits. Participants will be asked to maintain their normal daily activities.
  Interventions: Other: Usual Care
- Sub-study: Tele-prehabilitation and inspiratory muscle training program (Experimental): Eligible participants awaiting lung cancer surgery that have been randomised into the intervention arm will be re-randomised to receive either the STTARRS (larger trial) intervention or the STTARRS intervention PLUS an individualised inspiratory muscle training and walking program delivered by a physiotherapist using telehealth in the lead up to their lung cancer surgery.
  The inspiratory muscle training program includes an inspiratory muscle training explanatory video and an individually prescribed dosage and resistance for inspiratory muscle training and walking program, delivered via telehealth.
  Interventions: Behavioral: Tele-prehabilitation education session: Surgery School; Behavioral: Individualised Inspiratory Muscle Training and Walking Program
- Sub-study: Tele-prehabilitation intervention (Active Comparator): The Teleprehabilitaiton intervention (also known as Surgery School) is a one-off group based education session delivered online. Video presentations of 8-10 key prehabilitation education areas will be facilitated by a live clinician facilitator who will introduce the educational content and answer any questions. All standardised video presentations during the session will be made available to participants through an online password-protected video repository hosted on a video platform after the session and will be available until their surgery.
  Interventions: Behavioral: Tele-prehabilitation education session: Surgery School

INTERVENTIONS:
Behavioral: Tele-prehabilitation education session: Surgery School — Online telehealth education program using videos and a live clinician facilitator
  Arms: Sub-study: Tele-prehabilitation and inspiratory muscle training program; Sub-study: Tele-prehabilitation intervention; Tele-prehabilitation intervention (Intervention Group)
Behavioral: Individualised Inspiratory Muscle Training and Walking Program — An individualised inspiratory muscle training and walking program delivered by a Physiotherapist using telehealth.
  Arms: Sub-study: Tele-prehabilitation and inspiratory muscle training program
Other: Usual Care — Usual care alone. Usual care will be reviewed every four months during the trial and site leads will be asked to provide information about any changes to usual hospital and medical care at their site.
  Arms: Usual care alone (Control Group)

SUMMARY:
The physiological challenge of major surgery has been likened to running a marathon. In both cases, preparation is critical. Yet, many patients undergo major surgery without understanding the potential consequences.

The STTARRS trial aims to test the effect of an education program delivered via telehealth in people preparing for lung or major abdominal cancer surgery , compared with usual care on the development of a respiratory complications after surgery.

The secondary aims will be to determine the effect of the online education program for people preparing for lung or major abdominal cancer surgery compared to usual care on the following outcomes; acute hospital length of stay, surgical recovery, physical function and activity, self-efficacy, behaviour change, symptoms, health-related quality of life, number of days alive and out of hospital and health service usage and survival.

This trial includes one sub-study. The sub-study will recruit eligible people preparing for lung cancer surgery. In the sub-study, 35 participants will receive an individualised inspiratory muscle training and walking program delivered and monitored by telehealth in addition to the main STTARRS trial intervention before surgery.

ELIGIBILITY:
Inclusion Criteria:

* Preparing for lung cancer (open or video assisted) or major abdominal cancer surgery (e.g. upper GI, hepatobiliary or colorectal, open or video assisted).
* Provide consent
* Have primary treating surgeon approval
* Proficient in English to understand testing, video interventions as well as outcome assessments.

Exclusion Criteria:

* Concurrent, actively treated other malignancy or history of other malignancy treated within the past year.
* Severe or unstable psychiatric, cognitive or substance abuse disorders, such that precludes informed consent or interferes with cooperation with trial requirements or current inpatients.
* Current inpatients or incarcerated
* Surgery date booked <7 days from consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 515 (Estimated)
Dates: Start 2025-01-22 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Post operative Pulmonary Complication (PPC) | Daily for up to 7 days post operatively or until hospital discharge.
  Post operative pulmonary complications (PPC) will be assessed using the Melbourne Group Score (MGS). The MGS is an eight-item checklist. Minimum score 0, Maximum score 8. Participants are identifying as having a PPC if they score four or more in a 24-hour period.

SECONDARY OUTCOMES:
Diagnosis of pneumonia | Daily up to postoperative day 7 or until hospital discharge
  Diagnosis of pneumonia (Y/N) classified according the centre for disease control definition.
Postoperative complications | Postoperative day 3,5,10 unless discharge prior and 30 days post operative.
  Complications after surgery will be defined as any deviation from the normal postoperative course and classified according to the Clavien-Dindo classification. from Grade I through GradeV. Higher classifications indicating complications that require more complex interventions.
Number of days alive and out of hospital | 30 days, 6 months and 12 months post operative
  DAoH-30, DAoH-180, DAoH-365 (days alive and out of hospital 30, 180, 365 days post operatively): a patient centric metric and composite outcome that integrates several clinically important outcomes: hospital length of stay, re-admission or discharge to a destination other than origin (usually home) as well as survival. Higher numbers indicate a greater time alive and out of hospital post operatively.
Maximal Inspiratory Pressure (MIP) | Baseline and preoperatively at centres participating in the inspiratory muscle training sub study
  Maximal Inspiratory Pressure (cm H2O) will be assessed using a small handheld device using 3 tests of inspiratory muscle strength recording the highest value. Undertaken at centres participating in the sub study.
Physical activity levels - subjective | Baseline, Preoperatively, 30 days post operative
  Physical activity levels will be documented subjectively using the International Physical Activity Questionnaire - Short Form (IPAQ-SF). The IPAQ-SF is a questionnaire used internationally to obtain comparable estimates of physical activity. The questionnaire comprises seven questions related to physical activity at different levels of intensity and sitting time. Results will be reported in categories (low activity levels, moderate activity levels or high activity levels) and a continuous variable (MET minutes a week). Higher METs or categories indicate higher levels of physical activity.
Physical activity levels - objective | Baseline, Preoperatively, 30 days post operative
  Physical activity levels will be collected objectively using wearable monitors, such as fitbits for three days at baseline, three days after the intervention and at 30 days postoperatively. Physical activity variables will include the total number of daily steps, daily minutes of moderate to vigorous physical activity (MVPA), peak 1-minute cadence (the highest single minute of steps recorded), and peak 30-minute cadence (the average steps/min for the highest non-consecutive 30 minutes in a day). A minimum of 8 hours over 3 days is considered valid wear time for physical activity data. Values are described using mean +/- standard deviation and mean difference (MD) with 95% confidence intervals (95% CI).
Video and Surgery School Session Attendance (Intervention group only) | Preoperative timepoint
  Attendance at Surgery School session, length of time attended the Surgery School session and number of questions asked during Surgery School session.
Access to video outside the Surgery School Session (Intervention group only) | Preoperative timepoint
  The number of times the videos are accessed outside of the Surgery School session, site, day of week, time of day will be collected. Number of questions asked during Surgery School session.
Symptoms: electronic Edmonton Symptom Assessment System-revised ((e)ESAS-r) | Baseline (and repeated every 4 weeks for participants having treatment before surgery), Preoperative, Postoperative: 30 days.
  The electronic Edmonton Symptom Assessment System-revised ((e)ESAS-r) is a 10-item assessment tool for self-reporting symptom intensity via electronic platforms for digital use. The (e)ESAS-r allows participants to rate the severity of common symptoms as well as the opportunity to rate 'other problems' as nominated by the participant on a scale from 0 to 10 with higher score indicating higher severity of symptoms
Behaviour Change | Preoperative timepoint, at hospital discharge (+3 days)
  Behaviour change will be measured using a bespoke questionnaire: STTARRS behaviour change questionnaire (SBCQ) developed to assess patient action related to information (a) contained within the videos and surgery school session (intervention group) and (b) for usual care participants information provided to them through educational materials. This patient reported experience measure will measure responses to questions on a 5-point Likert scale (strongly disagree to strongly agree). Results will be presented descriptively. Higher responses on the likert scales indicates a higher agreement.
Self-efficacy: Patient Activation Measure | Baseline, preoperative timepoint, 30 days and 6 months postoperative.
  Patient Activation Measure (PAM) is a questionnaire assessing three key domains: knowledge, skills, confidence to understand self-management ability. The PAM is a 13-item survey scored on a 100 point scale, with 4 activation levels validated for across time measures and used world-wide. PAM Levels 1 and 2 indicate lower patient activation, while PAM levels 3 and 4 indicate higher patient activation.
Treatment Burden: Multimorbidity Treatment Burden Questionnaire (MTBQ) | Baseline, preoperative timepoint, 30 days postoperative
  Multimorbidity Treatment Burden Questionnaire (MTBQ) is a 13 item questionnaire that assesses the perception of the effort required to self-manage their medical conditions and the impact that this has on their wellbeing. The MTBQ has demonstrated good content and construct validity, reliability and responsiveness. The MTBQ is scored from 0-100 with higher scores indicating higher treatment burden which fall into four categories: no burden (score 0), low burden (score <10), medium burden (10-22) and high burden (>=22).
Viewer perceptions of the intervention (intervention group only) | Preoperative timepoint
  Viewer perceptions of the intervention including perceived personal relevance will be assessed using a previously published questionnaire. The questionnaire includes questions on four domains: helpfulness, believability, novelty, and relevance of information. A total of 7 questions all rate on 0-6 Likert scales from strongly disagree to strongly agree, with higher score indicating stronger agreement and an additional yes/no question asked regarding whether participants intend to change any behaviours.
Feasibility of the teleprehabilitation program: Proportion of eligible patients participating | Time Frame: Through study recruitment, up to 2.5 years
  Portion of eligible patients participating will be collected and reported as a percentage of all patients eligible for the trial.
Feasibility of the teleprehabilitation program: Representativeness | Time Frame: Through study recruitment, up to 2.5 years
  Representativeness relative to a wider group of eligible patients presented descriptively
Feasibility of the teleprehabilitation program: Referral rates | Time Frame: Through study recruitment, up to 2.5 years
  Actual teleprehabilitation referral rates as a % of total eligible to be referred
Feasibility of the teleprehabilitation program: reasons for declining | Time Frame: Through study recruitment, up to 2.5 years
  Reasons for declining will be reported descriptively.
Acceptability | Preoperative timepoint, at hospital discharge (+3 days), 30 days post operative
  Participants will be asked to complete a survey regarding trial acceptability. The survey questions will be based upon the Theoretical Framework of Acceptability. The framework comprises seven domains designed to assess acceptability elements: perceived effectiveness, self-efficacy, affective attitude, ethicality burden, intervention coherence and opportunity costs.
Fidelity (treatment delivery): Tele-prehabilitation education session duration | Through study data collection, up to 2.5 years
  Treatment delivery: using duration of education session provided (minutes).
Fidelity (treatment delivery): Number of videos accessed | Through study data collection, up to 2.5 years
  Treatment delivery: total number of videos accessed, presented descriptively and also by video title.
Fidelity (treatment delivery): Number of video views | Through study data collection, up to 2.5 years
  Treatment delivery: using number of videos viewed, results presented descriptively .
Fidelity (treatment delivery): Telehealth implementation process concordance with implementation protocol. | Through study data collection, up to 2.5 years
  Treatment delivery (centre level): using process concordance with implementation protocol.
Fidelity (treatment delivery): viewing time | Through study data collection, up to 2.5 years
  Treatment delivery: using the time of participant viewing (minutes).
Fidelity (treatment receipt): participant attendance at telehealth zoom meeting | Through study data collection, up to 2.5 years
  Treatment receipt: % of participants who attend a session once booked in
Fidelity (treatment receipt): number of questions | Through study data collection, up to 2.5 years
  Treatment receipt: the number of questions per session will be recorded.
Fidelity (treatment receipt): participant retention at follow up | Through study data collection, up to 2.5 years
  Treatment receipt: the number of participants attending follow up will be recorded (% of total participants).
Participant satisfaction: Australian Hospital Experience Question Set (AHPEQS) | 30 days post operative
  The Australian Hospital Patient Experience Question Set (AHPEQS) is a 12-item questionnaire (ten core items and two sub-items) used to measure patient satisfaction with recent treatment. Questions are measured on responses from always to never or didn't apply. Results will be reported descriptively with positive responses indicating greater satisfaction with recent treatment.
Health related quality of life: EORTC QLQ-C30 | Baseline, Preoperative, 30 days, 6 months and 12 months post operative
  European Organisation for the Research and Treatment of Cancer (EORTC QLQ- C30) core questionnaire is a measure composed of five multi-item domains (physical, role, emotional, cognitive function and social functioning). All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level. A high score for a functional scale represents a high/healthy level of functioning. A high score for the global health status / quality of life represents a high quality of life but a high score for a symptom scale / item represents a high level of symptomatology / problems. The EORTC QLQ-C30 Summary score will also be reported and is calculated from the mean of 13 of the 15 QLQ-C30 scale, with higher score indicating a higher quality of life. This tool has established validity and reliability in cancer.
Postoperative Quality of Recovery: Postoperative Quality of Recovery Score (PostopQRS) | Preoperative timepoint, 3 days and 6 days postoperatively (if not discharged prior), 30 days and 6 months postoperative
  The Postoperative Quality of Recovery Score (PostopQRS) is a multidimensional recovery assessment tool that is a verbal questionnaire. It has proven patient user acceptance and has been validated to be performed either face to face or over the telephone. The core domains include physiologic, nociceptive, functional, cognitive and emotional recovery and satisfaction with care, that is designed for use over multiple timepoints. The PostopQRS provides objective assessment of post-operative recovery, analysing the core domains of recovery, namely physiologic, nociceptive, functional, cognitive and emotional recovery compared to a unique individual preoperative baseline score. Recovery is then scored for each domain, and patients must recover in all tests within the domain to be scored as recovered. "All domains" recovery implies recovery in all of the five recovery domains.
Length of hospital stay | at hospital discharge
  Length of hospital stay will be documented from the medical records by a blinded assessor at each centre.
Health service use and costs | at hospital discharge, 30 days, 6 and 12 months post operative
  Captured in following ways:
  (i) hospital services and the use of health care services outside of hospital. (ii) Patients will be surveyed on their use of health services outside the hospital at 6 and 12 months postop follow-up using a questionnaire. (iii) Cost of program delivery
Exploratory Outcomes | through study completion, up to 3 years
  Teleprehabilitation is an intervention suitable for patients of low to moderately high perioperative risk levels, however subgroup analyses based on risk provide the opportunity to explore if teleprehabilitation offers additional benefits to patients of increasing risk level. Surgical procedure: Differences in PPC rates between the two surgical groups (abdominal and lung) and between those receiving or not receiving neo-adjuvant therapy before abdominal cancer surgery will be explored.

OTHER OUTCOMES:
Sex | Baseline
  After consent, participants' demographic data will be extracted from their medical record. Sex will be recorded as a categorical variable with categories: female, male, other.
Date of birth | Baseline
  After consent, participants' demographic data will be extracted from their medical record, including date of birth (years).
Height | Baseline
  After consent, participants' demographic data will be extracted from their medical record, including height (cm).
Weight | Baseline
  After consent, participants' demographic data will be extracted from their medical record, including weight (kg).
Primary language spoken | Baseline
  After consent, participants' demographic data will be extracted from their medical record, including primary language spoken (name of).
Proposed surgery | Baseline
  After consent, participants' clinical data will be extracted from their medical record, including proposed surgery (category of abdominal cancer or lung cancer surgery) and description of surgery.
Medical history | Baseline
  After consent, participants' clinical data will be extracted from their medical record, including medical conditions.
Social history: live alone | Baseline
  After consent, participants' social data will be extracted from their medical record, including living situation, living alone (yes/no).
Social history: partner | Baseline
  After consent, participants' social data will be extracted from their medical record, including living situation, if they have a partner (yes/no).
Work status | Baseline
  After consent, participants' demographic data will be extracted from their medical record, including work status.
Postcode | Baseline
  After consent, participants' demographic data will be extracted from their medical record, including postcode (zip code).
American Society of Anaesthesiologists (ASA) score | Baseline
  The American Society of Anaesthesiologists (ASA) score is a longstanding score that includes a subjective assessment of a patient's overall health according to five classes; (i) Patient is a completely healthy fit patient, (ii) Patient has mild systemic disease, (iii) Patient has severe systematic disease that is not incapacitating, (iii) Patient has severe systemic disease that is not incapacitating, (iv) Patient has incapacitating disease that is a constant threat to life or (v) A moribund patient who is not expected to live 24 hours with or without surgery. A higher category indicates higher risk.
Assess Respiratory Risk in Surgical Patients in Catalonia (ARISCAT) score | Baseline
  The Assess Respiratory Risk in Surgical Patients in Catalonia (ARISCAT) score is a valid tool for determining a patient's risk score for developing postoperative pulmonary complications. A higher score indicates higher risk of postoperative pulmonary complications and is classified as: low risk <26, intermediate risk: 26-44, and high risk : >=45.
Frailty | Baseline
  Frailty is a multidimensional geriatric syndrome characterised by a decline of physical and cognitive reserves that leads to increased vulnerability. It will be measured using the modified Reported Edmonton Frail Scale. The scale is a questionnaire with 13 items with a total score of 0 to 18. Scores are converted into the following categories: (0-5) not frail, (6-7) apparently vulnerable, (8-9) mild frailty, (10-11) moderate frailty and (12-18) severe frailty.
Survival | 12 months post operative
  Patients will be followed to assess if they are alive at 12 months post operatively.
Surgical and anaesthetic information | at hospital discharge
  Intraoperative details of surgical procedure, type of anaesthesia and reversal agent

CONTACTS AND LOCATIONS:
Overall Officials: Linda Denehy, B AppSc (Physio), PhD, Principal Investigator — University of Melbourne
Locations (6):
- Australia (6):
  - John Hunter Hospital, New Lambton Heights, New South Wales
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Launceston General Hospital, Launceston, Tasmania
  - Austin Health, Heidelberg, Victoria
  - Royal Melbourne Hospital, Melbourne, Victoria
  - Fiona Stanley Hospital, Perth, Western Australia

IPD SHARING:
Plan to Share IPD: No